CLINICAL TRIAL: NCT06054594
Title: Resistance Training and Cardiometabolic Risk in Women With Metabolically Healthy and Unhealthy Obesity
Brief Title: Resistance Training and Cardiometabolic Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec a Montréal (Other)
Responsible Party: Principal Investigator, Antony Karelis, Professor, Université du Québec a Montréal
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UQAM-SAP
Record Dates: First submitted 2023-09-12; First posted 2023-09-26 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Resistance Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metabolically healthy obesity (MHO) (Experimental): Healthy/normal metabolic profile
  Interventions: Other: Resistance exercise
- Metabolically unhealthy obesity (MUHO) (Experimental): Abnormal metabolic profile
  Interventions: Other: Resistance exercise

INTERVENTIONS:
Other: Resistance exercise — After baseline testing, participants followed a progressive resistance training program 3 times a week for 4 months.

SUMMARY:
Little is known on the effects of resistance training (RT) alone in individuals with metabolically healthy obesity (MHO) and metabolically unhealthy obesity (MUHO). The present study aimed to examine the impact of RT on body composition, physical performance, lipid-lipoprotein profile, inflammation, and glucose-insulin homeostasis in 51 sedentary, postmenopausal women categorized as MHO vs MUHO, according to the Karelis and Rabasa- Lhoret classification or a single-phenotype adiposopathy approach (the plasma adiponectin (A)/leptin (L) ratio). Participants followed a 4-month weekly RT program of 3 non-consecutive days of 6 exercises of major muscle groups (3 sets of 10 repetitions at 80% 1-RM).

DETAILED DESCRIPTION:
Several studies have examined MHO individuals' responses to weight loss interventions. Caloric restriction decreases body weight and body fat, notably visceral fat accumulation, of both MHO and MUHO pre- and postmenopausal women, although changes in MUHO women are usually more important. In addition, while insulin sensitivity of MUHO women increases after a 12-week diet, it is significantly worsened in postmenopausal MHO women. In this regard, previous works have shown discordant data of interventions including physical activity on the cardiometabolic risk and more particularly, insulin sensitivity. Indeed, diet or aerobic training alone or combined aerobic and resistance training (RT), in men and postmenopausal women yielded promising results as insulin sensitivity increased in both MUHO and MHO participants, with greater changes in the MUHO groups. However, the heterogeneity of the population (analysis without considering sex differences) as well as the type and duration (3 to 6 months) of different interventions make it difficult to generalize these results. As an example, insulin sensitivity was improved in MUHO men and women, while it remained unchanged in MHO participants after a 9-month intervention combining diet and exercise. Moreover, a 14-week community-based aerobic exercise program increased participants' cardiorespiratory fitness and reduced the number of metabolic syndrome components of MHO men and women. However, to the best of our knowledge, no study has compared yet the impact of a RT program on MUHO and MHO individuals.

ELIGIBILITY:
Inclusion criteria:

* cessation of menstruation for more than 1 year and a follicle-stimulating hormone level ≥ 30 IU/L
* sedentary for at least 3 months (< 2 h/week of structured exercise)
* non-smokers
* free of known inflammatory diseases
* no use of hormone replacement therapy
* body mass index ≥ 30 kg/m2
* low to moderate alcohol consumption (< 2 drinks/day)

Exclusion criteria:

* history of cardiovascular disease
* type 2 diabetes
* orthopedic limitations.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-01; Primary Completion 2011-06-09 (Actual); Study Completion 2011-06-09 (Actual)

PRIMARY OUTCOMES:
Insulin resistance (IR) | Baseline and after 4 months
  Homeostasis Model Assessment (HOMA)-IR index = insulin (μUI/mL) x glucose (mmol/L)/22.5

CONTACTS AND LOCATIONS:
Overall Officials: Antony Karelis, PhD, Principal Investigator — Université du Québec a Montréal

IPD SHARING:
Plan to Share IPD: No